CLINICAL TRIAL: NCT03149380
Title: Evaluating the Effectiveness of Web-based Education Via Alzheimer's Universe (Www.AlzU.Org) on Knowledge and Behavior: A Randomized Trial
Brief Title: Effectiveness of Alzheimer's Universe (Www.AlzU.Org) on Knowledge and Behavior
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: PI withdrawn
Sponsor: Weill Medical College of Cornell University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 1311014539
Record Dates: First submitted 2017-01-13; First posted 2017-05-11 (Actual); Last update posted 2023-03-22 (Actual); Status verified 2023-03

CONDITIONS: Alzheimer Disease; Alzheimer Disease, Late Onset; Memory Loss; Patient Education as Topic
MeSH Terms: conditions — Alzheimer Disease; Memory Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Subjects will be given access to educational content on AD using interactive learning strategies
  Interventions: Behavioral: Web-based education
- Time-neutral control (Sham Comparator): Subjects will be given access to time-neutral general educational content on AD
  Interventions: Behavioral: Web-based education

INTERVENTIONS:
Behavioral: Web-based education — The investigators will utilize interactive lessons and activities to educate about Alzheimer's disease prevention, treatment and caregiving, with focus on evidence-based lifestyle and nutritional recommendations that have been associated with delaying cognitive decline.

SUMMARY:
To evaluate the effectiveness of an online educational course on Alzheimer's disease (AD) prevention, treatment and caregiving.

DETAILED DESCRIPTION:
Alzheimer's Universe (www.AlzU.org) was created to provide online education about Alzheimer's disease (AD), with a focus on family members of people with AD, people with mild cognitive impairment due to AD and mild AD, caregivers, healthcare providers, medical students, college students and high school students. The website provides evidence-based courses with interactive lessons and activities that have been shown to increase knowledge about AD, willingness to participate in an AD prevention clinical trial, and intent to make specific lifestyle changes in effort to reduce AD risk.

ELIGIBILITY:
Inclusion Criteria:

* greater than or equal to 14 years old with a friend, family member or acquaintance with Alzheimer's disease or memory loss, OR a person diagnosed with mild memory loss (including mild cognitive impairment due to Alzheimer's disease or mild Alzheimer's disease), OR an AD caregiver, OR healthcare providers, OR a medical student, college student or high school student.

Exclusion Criteria:

* < 14 years old, OR diagnosis of moderate or severe Alzheimer's disease

Min Age: 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2017-01 (Estimated); Primary Completion 2023-12 (Estimated); Study Completion 2024-10 (Estimated)

PRIMARY OUTCOMES:
Knowledge of AD Preventative behaviors | 12 months
  Knowledge is calculated as a positive change on multiple-choice questions about AD between pre vs. post-completion of educational material
Willingness to Engage in AD Preventative behaviors | 12 months
  Willingness is calculated as a positive change on questionnaires evaluating AD-preventative behaviors between pre vs. post-completion of educational material

SECONDARY OUTCOMES:
Participant Satisfaction | 12 months
  The investigators will assess general satisfaction with the educational modules via pre vs post-intervention participant surveys
Behavioral Assessments | 12 months
  The investigators will evaluate related behavioral assessments via pre vs post-intervention participant surveys

CONTACTS AND LOCATIONS:
Overall Officials: Richard Isaacson, MD, Principal Investigator — Weill Medical College of Cornell University
Locations (1):
- Weill Medical College of Cornell University, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Direct hyperlink to Alzheimer's Universe website — http://www.AlzU.org/